CLINICAL TRIAL: NCT04962334
Title: Effect of Nutritional Formula Supplementation on Growth of Prepubertal Children Treated With Stimulants Medications for ADHD. A Randomized Double-blind, Placebo-controlled Trial
Brief Title: Effect of Nutritional Formula Supplementation on Growth of Prepubertal Children Treated With Stimulants Medications for Attention Deficit Hyperactivity Disorder (ADHD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: NG Solutions Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: rmc013521ctil
Record Dates: First submitted 2021-06-29; First posted 2021-07-14 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: ADHD - Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional Standardized Supplementation Formula (Experimental): Powder added to water, containing about 25% of recommended daily recommended intake (DRI) for calories, high protein (25% of calories) and multivitamin and mineral (25%-100% of DRI for recommended daily allowance (RDA) or adequate intake
  Interventions: Dietary Supplement: Nutritional supplementation standardized formula.
- Placebo (Placebo Comparator): Low caloric formula (Powder added to waster) without added vitamins and minerals
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nutritional supplementation standardized formula. — Powder added to water, containing about 25% of recommended daily recommended intake (DRI) for calories, high protein (25% of calories) and multivitamin and mineral (25%-100% of DRI for recommended daily allowance (RDA) or adequate intake
  Arms: Nutritional Standardized Supplementation Formula
Dietary Supplement: Placebo — Low caloric formula (powder added to water) without added vitamins and minerals
  Arms: Placebo

SUMMARY:
The proposed study is a double blind, randomized, placebo controlled study. The aim of the study is to evaluate the effect of nutritional formula supplementation on growth of prepubertal children treated with stimulants medications of ADHD.

70 Participants treated with stimulants medications of ADHD will be randomly assigned either to the intervention group or the placebo control group. Randomization for the two study groups will be made in a ratio of 1:1. Both participants and study team will be blinded to the type of treatment that each patient will receive during the study. Randomization will be stratified according to gender.

Participants in the intervention groups will be treated with the study formula and participants in the control group will be treated with a placebo low caloric formula (Powder added to water). The study will continue for 6 months of intervention versus active placebo, with additional 6 months (an extension period), in which participants at both groups, the intervention and the placebo, will be offered to continue their participation in the study with the active study supplement.

In addition, 30 prepubertal healthy siblings will be recruited to the study in order to compare baseline eating and physical activity patterns of ADHD children treated with stimulants to their healthy untreated siblings at the same age range. Participants' siblings will only complete once the nutritional and physical activity questionnaire and report height and weight measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Boys aged ≤ 10 years and girls aged ≤ 9 years.
2. Children treated with stimulants medications for ADHD for at list 3 months.
3. Prepubertal -Tanner stage 1 (gonadarche) (boys: testicular volume < 4, girls: breast at Tanner stage 1)
4. Normal weight status: BMI-SDS ≤ 85th percentile for age and gender according to the CDC 2000 growth charts
5. Signing inform consent forms

Exclusion Criteria:

1. Diagnosis of GH Deficiency or treatment with GH
2. Any known chronic disease or dysmorphic syndrome including bone diseases, organic brain diseases, neurological disease, past or current malignancy, chronic cardiac, renal or pulmonary problems
3. Any known gastrointestinal disease including malabsorption
4. Any known organic reason for growth retardation
5. Milk allergy.
6. Any chronic treatment with additional medication beside stimulants that might affect appetite, weight, or growth (for example SSRI's).

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
height standard deviation score (SDS) | at 6 months
weight standard deviation score | at 6 months

SECONDARY OUTCOMES:
BMI SDS | at 6 months
Fat Mass | at 6 months
Lean body mass | at 6 months
Muscle mass | at 6 months
Change in dietary patterns measured by Child Eating Behaviour Questionnaire | At 6 months
Change in ADHD symptoms measured by Vanderblit ADHD Parent Rating Scale | at 6 months
Change in physical activity patterns measured by physical activity questionnaire | at 6 months

OTHER OUTCOMES:
height SDS | at 12 months
Weight SDS | at 12 months
BMI SDS | at 12 months
Fat mass | at 12 months
Lean body mass | at 12 months
Muscle mass | at 12 months
Change in dietary patterns measured by Child Eating Behaviour Questionnaire | at 12 months
Change in ADHD symptoms measured by Vanderblit ADHD Parent Rating Scale | at 12 months
Change in physical activity measured by physical activity questionnaire | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof, Principal Investigator — Schneider Children's Medical Center
Locations (1):
- Schneider children's medical center, Petah Tikva, Israel